CLINICAL TRIAL: NCT03146884
Title: Swiss Autoimmune Hepatitis Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Fondazione Epatocentro Ticino (Other)
Responsible Party: Sponsor
Other Study IDs: SASL38 - Swiss AIH Cohort
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2025-08-18 (Actual); Status verified 2025-08

CONDITIONS: Hepatitis, Autoimmune; Autoimmune Hepatitis
Keywords: Autoimmune Hepatitis; AIH; Cohort
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — 1. Serum (BD Vacutainer® SST II Advance)
  2. RNA (PAXgene™ Blood RNA tube- 762165)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Research project in which biological material is sampled and health-related personal data is further used and collected.

Coded data are used.

DETAILED DESCRIPTION:
To collect high quality prospective data on a rare disease in order to elucidate epidemiology, natural history, response to treatment and outcome. In addition, a biobank allows addressing specific scientific issues on a variety of open questions. The cohort will provide a platform for carrying out scientific research projects on AIH. In addition, the cohort will allow collaborations with reference networks on AIH abroad.

Measurements and procedures: Enrolment visit and one follow-up visit at least once a year are planned. An additional follow-up visit at 6 months postdiagnosis is planned for newly diagnosed patients.

Whole blood is collected for biobanking once a year Optionally, if available and collected during normal clinical procedures, liver fragments are obtained.

Number of subjects projected for the entire study (all sites combined): 500 (corresponding to 1/3 of the estimated global AIH population residing in Switzerland, assuming a disease prevalence of 20:100,000)

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of AIH, either type I or type II
* Only patients living in Switzerland

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with AIH, either type I or type II living in Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease course | 3 years
  Observing disease course
Disease features | 3 years
  Observing disease features in Swiss population and see if they are similar to other countries'
Response to treatment | 3 years
  Observing response to treatment
Overall survival | 3 years
  Observing overall survival
Transplantation-free survival rate | 3 years
  Observing transplantation-free survival rate

CONTACTS AND LOCATIONS:
Locations (20):
- Switzerland (20):
  - Fondazione Epatocentro Ticino, Lugano, Canton Ticino
  - Gastroenterologie und Hepatologie Clarunis - Universitäres Bauchzentrum, Universitätsspital Basel, Basel
  - Universitäts-Kinderspital beider Basel UKBB, Gastroenterologie&Ernährung, Basel
  - Inselspital, Bern
  - Kinderklinik, INSELSpital, Universität Bern, Pädiatrische Gastroenterologie, Hepatologie und Ernährung, Bern
  - Kantonsspital Graubünden, Chur
  - Hôpitaux Universitaires de Genève, Centre Suisse des Maladies du foie de l'Enfant- Département de l'Enfant et de l'Adolescent, Geneva
  - Hôpitaux Universitaires de Genève, Service de Gastroentérologie & Hépatologie, Département des Spécialités, Geneva
  - CHUV: Centre hospitalier universitaire vaudois, Lausanne
  - CHUV Département femme-mère-enfant, Lausanne
  - Kantonsspital Baselland, Liestal
  - Kinderspital Luzern LUKS, Pädiatrische Gastroenterologie, Lucerne
  - Luzerner Kantonsspital, Lucerne
  - EOC Ospedale Regionale di Lugano - Italiano, Lugano
  - Ostschweizer Kinderspital, Sankt Gallen
  - Kantonsspital St.Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Kinderspital Winterthur, Klinik für Gastroenterologie & Hepatologie, Winterthur
  - Universitäts-Kinderspital Zürich - Eleonorenstiftung, Zurich
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No